CLINICAL TRIAL: NCT02003703
Title: Comparative Efficacy of an Intensified Re-vaccination Scheme for Hepatitis B Virus Infection Among Patients Infected With HIV : A Randomised Trial
Brief Title: Comparative Efficacy of an Intensified Re-vaccination Scheme for Hepatitis B Virus Infection Among Patients Infected With HIV .
Acronym: CORE-HIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Roche Pharma AG (Industry); GlaxoSmithKline (Industry); Aclin Laboratory (Other)
Responsible Party: Principal Investigator, Felipe Martinez, MD, Universidad de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 45/2012
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis B; HIV
Keywords: Vaccine; Primary Prevention; Immunogenicity
MeSH Terms: conditions — Hepatitis B | interventions — Engerix-B; halofantrine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recombinant Hepatitis B Virus Vaccine (High Dose) (Experimental): Patients allocated to this arm will receive three doses of 40mcg each of recombinant hepatitis B vaccine (Engerix-B (R)). Doses will be administered at 0, 1 and 2 months.
  Interventions: Biological: Recombinant Hepatitis B Virus Vaccine
- Recombinant Hepatitis B Virus Vaccine (Standard Dose) (Active Comparator): Patients allocated to this arm will receive three doses of 20mcg each of recombinant hepatitis B vaccine (Engerix-B (R)). Doses will be administered at 0, 1 and 2 months.
  Interventions: Biological: Recombinant Hepatitis B Virus Vaccine

INTERVENTIONS:
Biological: Recombinant Hepatitis B Virus Vaccine
  Other Names: Engerix B (GlaxoSmithKline)

SUMMARY:
Hepatitis B virus infection is a common occurrence among patients with HIV. Effective vaccines are available, but there's some uncertainty regarding specific dosages, specially among those who have not responded to an initial vaccination. The purpose of this study is to determine the effectiveness of a simplified immunization schedule compared to a high-dose one.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age.
* Patients infected with Human Immunodeficiency Virus (HIV)
* Failed previous vaccination with a standard dose scheme of recombinant hepatitis B vaccine (20mcg at 0, 1 and 6 months). Nonresponders will be considered as those patients presenting a hepatitis B surface antigen antibody titer lower than 10UI/mL 4 to 8 weeks after the last dose of the vaccine.
* Provision of informed consent.

Exclusion Criteria:

* Proven Hepatitis B virus infection (acute or chronic).
* Proven hypersensitivity to the vaccine or any of its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-05; Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Serologic Response | 4-8 weeks After Exposure
  Number of participants with positive hepatitis B surface antigen (HBsAg) antibodies 4 to 8 weeks after completion of the vaccination schemes.

SECONDARY OUTCOMES:
Local Reactions to Vaccine | One Week after Exposure
  Number of participants presenting dermatologic reactions to the vaccine up to one week after exposure.
Systemic Reactions to the Vaccine | One Week after Exposure
  Number of participants presenting any systemic adverse reaction attributable to vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Fuster, MD, Principal Investigator — Hospital Gustavo Fricke, Viña del Mar, Chile; Jose I Vargas, MD, Principal Investigator — Escuela de Medicina, Universidad de Valparaíso, Chile; Daniela Jensen, MD, Principal Investigator — Escuela de Medicina, Universidad de Valparaíso; Felipe T Martinez, MD, Principal Investigator — Centro de Investigaciones Biomédicas, Escuela de Medicina, Universidad de Valparaíso
Locations (1):
- Hospital Gustavo Fricke, Viña del Mar, Región de Valparaíso, Chile

REFERENCES:
- [Derived] Vargas JI, Jensen D, Martinez F, Sarmiento V, Peirano F, Acuna P, Provoste F, Bustos V, Cornejo F, Fuster A, Acuna M, Fuster F, Soto S, Estay D, Jensen W, Ahumada R, Arab JP, Soza A, Fuster F. Comparative Efficacy of a High-Dose vs Standard-Dose Hepatitis B Revaccination Schedule Among Patients With HIV: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2120929. doi: 10.1001/jamanetworkopen.2021.20929. PMID 34424307